CLINICAL TRIAL: NCT02549378
Title: Study of the Impact of Changes in Carbonemia on Microcirculation in Patients - A Monocentric Study
Brief Title: Study of the Impact of Changes in Carbonemia on Microcirculation in Patients Achieving a Test Hypercapnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1308031
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Microcirculation; Blood Circulation
Keywords: microcirculation; confocal microscopy; hypocapnia
MeSH Terms: conditions — Hypocapnia | interventions — Microscopy, Confocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with a hypercapnia test (Experimental): confocal microscopy patients with a hypercapnia test
  Interventions: Device: confocal microscopy

INTERVENTIONS:
Device: confocal microscopy — microvessel diameter measured by confocal microscopy

SUMMARY:
The microcirculatory alterations is common in circulatory failure, especially during sepsis. The severity of these changes and their sustainability are responsible of multi organ failure and ultimately death. The optimization of microcirculatory flow could be a central objective of the management of patients hospitalized in intensive care.

Microcirculation includes all blood vessels of a diameter smaller than 100 micrometer. It represents the largest heat exchange surface of the body and is involved in tissue oxygenation. Microcirculatory flow is conditioned by the macrocirculation (heart rate and blood pressure) and the state of the microcirculation (thrombosis, vasoconstriction ...). The role of the CO2 in regulating microcirculatory flow is little studied. A recent work of our team and the oldest work in the literature lead to believe that CO2 has a specific role in modulating microcirculatory flow. No study to date precisely studied the impact of changes in the microcirculatory flow carbonemia .

The hypocapnia test is carried out in a standardized manner by inhalation of a mixture enriched in CO2 7% allows a significant increase in carbonemia. Hypocapnia will in turn obtained by a calibrated voluntary hyperventilation test.

Direct visualization of microcirculation by confocal microscopy is now considered the gold standard for exploring the microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* patients from achieving hypercapnia test the CHU of Saint-Etienne
* non smoking
* non diabetic
* affiliated with or entitled to a social security system
* Written consent

Exclusion Criteria:

* subjects not performing the test hypercapnia in full
* patients with dermatological pathology at the study area
* patient with Raynaud's syndrome
* Patients with known bleeding disorders
* refusal to consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
microcirculatory flow (cells / min) measured by confocal microscopy | Day1
  microcirculatory flow (cells / min) measured by confocal microscopy in hypocapnic patients

SECONDARY OUTCOMES:
microvessel diameter (micrometer) measured by confocal microscopy | Day1
  microvessel diameter (micrometer) measured by confocal microscopy in hypocapnic patients

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Gergelé, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France